CLINICAL TRIAL: NCT01221181
Title: Eculizumab Therapy for Dense Deposit Disease and C3 Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Gerald B. Appel, Professor of Clinical Medicine, Nephrology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF2403
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dense Deposit Disease; Membranoproliferative Glomerulonephritis
Keywords: Dense deposit disease; C3 nephropathy; Eculizumab
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eculizumab (Experimental): Patients will receive Eculizumab and be observed for 60 minutes after the first 5 infusions, then 30 minutes after all subsequent infusions. Patients will not be allowed to take other immunomodulatory therapies during the study period but will continue on their other non-immunomodulatory therapies (e.g. ACE inhibitors, -statins, aspirin) without modifications unless clinically indicated. All patients, if unvaccinated, will be given N. meningitides vaccine at least two weeks prior to first eculizumab exposure. All female patients of childbearing potential will be asked to use adequate contraception methods during treatment and up to 5 months following discontinuation of eculizumab treatment.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Dosage/Frequency: 900 mg IV once a week for 4 weeks, 1200 mg IV week 5, then 1200 mg IV every 2 weeks through week 53.
  Other Names: Eculizumab (Soliris®)

SUMMARY:
This open label, non-blinded, proof of concept efficacy and safety study of eculizumab in patients with biopsy proven DDD or C3 nephropathy. The trial will consist of adult patients with these diseases who have > 1 gram of proteinuria or a decreased glomerular filtration rate (GFR), both predictors of a poor long-term outcome in many glomerular diseases. The patients will be treated with eculizumab for one year.

The goals will be to determine whether treatment leads to an improvement in kidney function, defined by remissions of proteinuria and improvements in estimated GFR (measured by serum creatinine), and to improvement in histologic parameters, including percentage of non-affected glomeruli, interstitial fibrosis, intensity of C3 staining of immunofluorescence, and amount of electron dense deposits by electron microscopy.

DETAILED DESCRIPTION:
Dense deposit disease (DDD), also called membranoproliferative glomerulonephritis (MPGN) type II, is a rare form of glomerulonephritis named because of the characteristic appearance of electron-dense material in the glomerular basement membrane observed on kidney biopsy. The principle immune defect in DDD is excessive activation of the alternative complement pathway, with deposition of complement components in the glomerular basement membrane. Hence, by immunofluorescence microscopy, there is heavy C3 deposited along the basement membrane. Some patients have been found to have deficiencies of Factor H or Factor I, inhibitors of C3 activation. Others have a C3 nephritic factor, an antibody that activates the alternative complement cascade. It has recently been recognized that C3 nephropathy, a rare glomerular disease with mesangial cell proliferation and C3 deposition by immunofluorescence microscopy, is associated with similar over-activation of the alternative complete cascade.

While DDD affects mostly children and young adults, in the series of 32 patients from Columbia with DDD whose biopsies were read from 1977-2007, 18 patients (56%) were older than 16 years of age at the time of diagnosis, and about 40% of patients were over 30 years old. The age division is important for two reasons. First, in the Columbia series, children appeared to have better clinical outcomes than adults. While 25.9% of all patients had a complete remission, there was a significant distinction between adults, of whom only 7.1% achieved complete remission, and children, of whom 46.1% achieved complete remission. Of the remaining patients who did not achieve remission, 42.9% of adults, compared to only 7.7% of children, progressed to end stage renal disease (ESRD) over a mean follow-up of over 5 years. Second, as there are no large clinical trials to guide specific interventions for DDD and the role of immunomodulatory therapies still remains controversial, many nephrologists advocate using immunomodulatory therapy only in selected adult patients.

Immunomodulatory therapies not specifically targeted to DDD, such as corticosteroids, cyclophosphamide, and calcineurin inhibitors, have either been unsuccessful or not studied in a meaningful number of patients to warrant routine use. However, as the principal defect underlying DDD is excessive activation of the alternative complement pathway, with deposition of complement components in the glomerular basement membrane, a therapy that directly targets the alternative complement pathway may prove particularly beneficial for this disease.

Eculizumab is a humanized monoclonal antibody that binds with high affinity to C5. The drug is FDA-approved for the treatment of paroxysmal nocturnal hemoglobinuria (in which mutations of complement regulatory proteins on hematopoietic cells lead to alternative complement pathway-mediated hemolysis). It is currently being studied for use in atypical hemolytic uremic syndrome, a rare disease marked by diffuse micro-thromboses related to activation of the alternative complement system. Eculizumab prevents cleavage of C5, thereby precluding formation of C5a, which has been implicated in glomerular inflammation in animal models of DDD. Moreover, by inhibiting the activation of C5, it prevents the formation of the membrane attack complex C5-9. Speculatively, this drug could provide effective, targeted therapy for patients with DDD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with biopsy proven DDD or C3 nephropathy, at least 18 years of age
* 24-hour urine protein > 1000 mg/day, urine protein:creatinine ratio > 1.0, or acute renal failure (defined as > 50% increase in serum creatinine from baseline)
* Willing and able to sign informed consent
* Patients of childbearing age must agree to use birth control
* Patients must be willing to be vaccinated against meningococcal disease or have documentation of previous vaccination against meningococcal disease

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable to sign informed consent
* Patients having received rituximab or another monoclonal antibody within 6 months of the trial
* Patients currently taking and unable to discontinue other immunomodulatory therapies (e.g. cyclosporine, high-dose steroids, mycophenolate mofetil) unless these other therapies are indicated for prophylaxis of transplant rejection (e.g. stable doses of mycophenolate mofetil and/or calcineurin inhibitor). Patients on chronic steroid therapy who are unable to taper down to <10 mg/day will be excluded.
* Patients of childbearing age who refuse to use birth control
* Patients with a baseline estimated GFR less than 30 ml/min/1.73m2
* Patients with other renal diseases (e.g. diabetic nephropathy, renal vascular disease) that would interfere with interpretation of the study.
* Patients with comorbid conditions that would interfere with completion of the trial (malignancies, congestive heart failure (CHF), recent myocardial infarction).
* Patients with known contraindications to the use of eculizumab, including refusal to receive N. meningitides vaccine prior to therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald B Appel, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, Glomerular Center, New York, New York
  - Columbia University Medical Center, Nephrology Clinical Research Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bomback AS, Smith RJ, Barile GR, Zhang Y, Heher EC, Herlitz L, Stokes MB, Markowitz GS, D'Agati VD, Canetta PA, Radhakrishnan J, Appel GB. Eculizumab for dense deposit disease and C3 glomerulonephritis. Clin J Am Soc Nephrol. 2012 May;7(5):748-56. doi: 10.2215/CJN.12901211. Epub 2012 Mar 8. PMID 22403278
- See also: Eculizumab for dense deposit disease and C3 glomerulonephritis — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3338285/
- See also: Pathology after eculizumab in dense deposit disease and C3 glomerulonephritis — http://www.ncbi.nlm.nih.gov/pubmed/22677550

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: Patients will receive Eculizumab and be observed for 60 minutes after the first 5 infusions, then 30 minutes after all subsequent infusions.
Period: Overall Study
Arm/Group | Eculizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 23.5 [20 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (NIH/OMB) Not Hispanic or Latino
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 6
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Creatinine [Median (Full Range); unit: mg/dl] | 1.75 [1.2 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Change in Proteinuria or Serum Creatinine Over Treatment Period
Description: This is designed to measure response to eculizumab through clinical and histological data, including a reduction in serum creatinine or in proteinuria, or histopathologic improvement. Any reduction in serum creatinine and/or proteinuria was included in our descriptive analysis.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Groups:
- Eculizumab: Eculizumab 900 mg IV one a week for 4 weeks, 1200 mg IV week 5, then 1200 mg IV every 2 weeks through week 53.
  Eculizumab: 900 mg IV once a week x 4 weeks, 1200 mg IV week 5, then 1200 mg IV every 2 weeks through week 53.
  Patients will be observed for 60 minutes after the first 5 infusions, then 30 minutes after all subsequent infusions. Patients will not be allowed to take other immunomodulatory therapies during the study period but will continue on their other non-immunomodulatory therapies (e.g. ACE inhibitors, -statins, aspirin) without modifications unless clinically indicated. All patients, if unvaccinated, will be given N. meningitidis vaccine at least two weeks prior to first eculizumab exposure. All female patients of childbearing potential will be asked to use adequate contraception methods during treatment and up to 5 months following discontinuation of eculizumab treatment.
Arm/Group | Eculizumab
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes